CLINICAL TRIAL: NCT03602508
Title: Treatment Persistence Among Patients With Overactive Bladder: A Retrospective Secondary Data Analysis in Asia Oceania
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 178-MA-3147
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2019-10

CONDITIONS: Overactive Bladder (OAB)
Keywords: darifenacin; fesoterodine; trospium; solifenacin; oxybutynin; tolterodine; Betmiga; YM178; mirabegron; Overactive bladder; propiverine; antimuscarinics; OAB; imidafenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron; Solifenacin Succinate; darifenacin; imidafenacin; Tolterodine Tartrate; oxybutynin; trospium chloride; fesoterodine; propiverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mirabegron: Patients on mirabegron as prescribed by a physician in routine clinical practice.
  Interventions: Drug: mirabegron
- antimuscarinics: Patients on one of the following antimuscarinics: solifenacin, darifenacin, imidafenacin, tolterodine, oxybutynin, trospium, fesoterodine or propiverine as prescribed by a physician in routine clinical practice.
  Interventions: Drug: solifenacin; Drug: darifenacin; Drug: imidafenacin; Drug: tolterodine; Drug: oxybutynin; Drug: trospium; Drug: fesoterodine; Drug: propiverine

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178; Betmiga
  Groups: mirabegron
Drug: solifenacin — oral
  Other Names: YM905; Vesicare
  Groups: antimuscarinics
Drug: darifenacin — oral
  Groups: antimuscarinics
Drug: imidafenacin — oral
  Groups: antimuscarinics
Drug: tolterodine — oral
  Groups: antimuscarinics
Drug: oxybutynin — oral
  Groups: antimuscarinics
Drug: trospium — oral
  Groups: antimuscarinics
Drug: fesoterodine — oral
  Groups: antimuscarinics
Drug: propiverine — oral
  Groups: antimuscarinics

SUMMARY:
The purpose of this study is to descriptively evaluate the persistence among adults treated with mirabegron or antimuscarinics in Australia, South Korea and Taiwan.

This study will also assess the persistence to the overall Overactive bladder (OAB) treatments of a patient, regardless of treatment discontinuation or switch to other OAB medications.

DETAILED DESCRIPTION:
This study is entirely descriptive using secondary medical claim and pharmacy prescription data. No formal comparisons between users of mirabegron and antimuscarinic will be made. Furthermore, no a priori hypothesis testing is intended.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a new prescription of the index medication within the index period;
* Patient received orally administered monotherapy for OAB on index date.

Exclusion Criteria:

* Patient with prior dispensing record of the index medication during the pre-index period;
* Patient received onabotulinumtoxin A and/or surgical intervention as part of the OAB treatment between the pre index and post-index period;
* Patient diagnosed with stress incontinence (International Classification of Diseases-10 (ICD-10) N39.3 or equivalent) or had dispensing record of medication for stress incontinence (duloxetine) before index date;
* Patient with urinary tract infection (ICD-10 N30.0 or equivalent) (for National Health Insurance Research Database (NHIRD) and Health Insurance Review and Assessment (HIRA) database) or a co-prescription of any antibiotics (for NostraData) on index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (aged ≥18 years; except for Taiwan ≥20 years old) with overactive bladder who received pharmacological treatment between 1st July 2015 and 29th February 2016.
Sampling Method: Non-Probability Sample
Enrollment: 5589 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Patients persistence to the index medication | Up to 12 months
  Persistence to the index medication (i.e. mirabegron; solifenacin; darifenacin; imidafenacin; tolterodine; oxybutynin; trospium; fesoterodine; propiverine) is defined as the time to discontinuation during the 1 year post-index period. Days with the index medication for each patient will be calculated as the sum of days of supply per prescription.

SECONDARY OUTCOMES:
Patients persistence to the overall Overactive Bladder (OAB) treatment regardless of treatment switching to other OAB medications | Up to 12 months
  Time to discontinuation of the overall OAB treatment during the one-year post-index period (persistence) is defined as days with the index medication (i.e. mirabegron; solifenacin; darifenacin; imidafenacin; tolterodine; oxybutynin; trospium; fesoterodine; propiverine) for each patient and days' supply of any OAB medication will be added up until the grace period exceeds 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Singapore Pte. Ltd.
Locations (2):
- Site AU10000, Sydney, Australia
- Site KR82001, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.